CLINICAL TRIAL: NCT00010192
Title: A Phase I Trial Of Rituximab And Interleukin-2
Brief Title: Rituximab Plus Interleukin-2 in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01404; 0037; CDR0000068454; OSU-0037; NCI-130; OSU-00H0223; U01CA076576 (NIH)
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; aldesleukin; Interleukin-2

ARMS (1):
- Treatment (rituximab and aldesleukin) (Experimental): Patients receive rituximab IV on days 1, 8, 15, and 22. Patients then receive low-dose aldesleukin SC on days 29-39, 43-53, 57-67, and 71-81, and intermediate-dose aldesleukin SC on days 40-42, 54-56, 68-70, and 82-84.
  Interventions: Biological: rituximab; Biological: aldesleukin; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Combining rituximab with interleukin-2 may kill more cancer cells. Phase I trial to study the effectiveness of rituximab plus interleukin-2 in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: Determine the dose-limiting toxicity of rituximab followed by low-dose and intermediate-dose pulse interleukin-2 (IL-2) in patients with CD20-positive B-cell lymphoid malignancy.

Determine the maximum tolerated dose of intermediate-dose pulse IL-2 in this patient population.

Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation study of intermediate-dose pulse aldesleukin.

Patients receive rituximab IV on days 1, 8, 15, and 22. Patients then receive low-dose aldesleukin subcutaneously (SC) on days 29-39, 43-53, 57-67, and 71-81, and intermediate-dose aldesleukin SC on days 40-42, 54-56, 68-70, and 82-84. Cohorts of 3-6 patients receive escalating doses of intermediate-dose pulse aldesleukin until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or immunophenotypically proven CD20-positive B-cell lymphoproliferative disorder

  * Recurrent or progressive low-grade B-cell lymphoma with at least one prior chemotherapy regimen (may have included monoclonal antibody)
  * Relapsed intermediate-grade or high-grade B-cell lymphoma or B-lineage acute lymphoblastic leukemia and patient not a candidate for, refused, or failed prior hematopoietic stem cell transplantation
* No chronic lymphocytic leukemia or lymphoma with more than 5,000/mm3circulating lymphoma cells
* Measurable or evaluable disease
* Must have failed standard curative therapy
* No CNS or leptomeningeal metastasis
* Performance status - Karnofsky 70-100%
* Performance status - ECOG 0-1
* At least 4 months
* Absolute neutrophil count at least 1,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)
* Platelet count at least 50,000/mm^3
* AST no greater than upper limit of normal (ULN)
* Bilirubin no greater than 1.5 times ULN
* Hepatitis B surface antigen negative
* Creatinine no greater than ULN
* No prior unstable coronary artery disease
* No New York Heart Association class III or IV congestive heart failure
* DLCO and FEV1 at least 50% of predicted
* HIV negative
* No other concurrent malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No infection requiring IV antibiotic therapy within the past 4 weeks
* No other major illness that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* See Disease Characteristics
* Prior antibody therapy allowed
* Prior interleukin-2 or interferon alfa allowed
* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior systemic corticosteroids
* At least 4 weeks since prior radiotherapy
* At least 4 weeks since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-12; Primary Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose preceding that at which at least 2 of 6 patients experience DLT using NCI CTC version 2.0 | 2 weeks
  Data collected will be descriptive and provide limited estimates of variability given the small sample sizes at each dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Porcu, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States